CLINICAL TRIAL: NCT00138918
Title: A Phase II Study of OGX-011 Given Prior to Radical Prostatectomy in Patients With Localized Prostate Cancer
Brief Title: Study of OGX-011 Given Prior to Radical Prostatectomy in Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R04-0092
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Clusterin; Neoadjuvant; Phase II
MeSH Terms: conditions — Prostatic Neoplasms | interventions — OGX-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: OGX-011 — See Detailed Description, Treatment Plan

SUMMARY:
The purpose of this trial is to assess the effects of combined therapy with androgen ablation and OGX-011 (an antisense to clusterin) given prior to radical prostatectomy on pathologic complete response rates in men with localized prostate cancer and high risk features.

DETAILED DESCRIPTION:
Clusterin as an anti-apoptotic cytoprotective chaperone protein upregulated in an adaptive cell survival manner that confers resistance to various cell death triggers, including hormone-, radiation-, and chemotherapy. In pre-clinical models, inhibition of clusterin expression using the second generation antisense OGX-011 can enhance cell death following treatment with androgen ablation, radiotherapy, and chemotherapy. In phase I clinical trials, OGX-011 has been well tolerated and a biologically effective dose has been identified in humans.

Study Design

This is an open-label, non-blinded, phase II clinical, tissue pharmacokinetic and pharmacodynamic study of weekly OGX-011 and neoadjuvant hormone therapy prior to radical prostatectomy in patients with localized prostate carcinoma and high-risk features.

Study Objectives

Primary Objectives

* To assess the effects of combined neoadjuvant hormone therapy (NHT) and OGX-011 prior to radical prostatectomy on pathologic complete response rates in men with high risk localized prostate cancer.

Secondary Objectives

* To quantify changes in clusterin expression in residual prostate cancer after treatment with NHT and OGX-011.
* To measure levels of full length OGX-011 in prostate tissues after 3 months of NHT.
* To assess the safety and tolerability toxicity of 3 months of OGX-011 and NHT prior to radical prostatectomy.
* To measure evidence of OGX-011's effect on clusterin expression in patient peripheral blood mononuclear cells (PBMNC).
* To measure evidence of OGX-011's effect on patient clusterin serum levels.
* To assess the effects of combined NHT and OGX-011 on time to PSA nadir.
* To determine PSA recurrence rates after combined NHT and OGX-011.

Key Eligibility Criteria

1. Histologically confirmed adenocarcinoma of the prostate, previously untreated
2. Potential candidate for radical prostatectomy
3. Any one of the following criteria (minimum of 2 positive biopsies):

   * Clinical stage T3
   * Serum PSA > 10 ng/ml
   * Gleason score 7-10
   * Gleason score 6 and > 3 positive biopsies
4. ECOG performance status 0-1
5. WBC ≥ 3.0 x 10^9/L
6. Hemoglobin ≥ 100 g/L
7. Platelets ≥ 100 x 10^9/L
8. PTT, INR, AST, ALT, creatinine, total bilirubin within normal limits

Treatment Plan

Approximately 45 newly diagnosed, previously untreated patients with clinically localized, high-risk prostate carcinoma will be entered into this trial. These patients will receive neoadjuvant hormone therapy (buserelin 9.9 mg subcutaneously x 1 injection with flutamide 250 mg orally T.I.D. for the first 4 weeks only) for 12 weeks in combination with OGX-011 (a 2'MOE phosphorothioate clusterin antisense oligonucleotide) weekly on a 4 week cycle for 3 courses. For week one, cycle one only, OGX-011 will be given on Days 1, 3 and 5. OGX-011 is given at a dose of 640 mg by intravenous infusion over 2 hours. Radical prostatectomy will take place within 14 days of the last dose of OGX-011.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate, previously untreated
2. Males ≥ 18 years of age.
3. Potential candidate for radical prostatectomy
4. Any of the following (minimum of 2 positive biopsies):

   * Clinical stage T3
   * Serum PSA > 10 ng/ml
   * Gleason score 7-10
   * Gleason score 6 and > 3 positive biopsies
5. ECOG performance status 0-1
6. WBC ≥ 3.0 x 10^9/L
7. Hemoglobin ≥ 100 g/L
8. Platelets ≥ 100 x 10^9/L
9. PTT, INR, AST, ALT, creatinine, total bilirubin within normal limits
10. Patients must sign an informed consent that complies with US Regulations (US 21 Code of Federal Regulations [CFR]) and the International Conference on Harmonization (ICH) Guideline for Good Clinical Practice (GCP) prior to undergoing treatment.

Exclusion Criteria:

1. Prior hormone, radiation, or chemotherapy for prostate cancer
2. Evidence of active infection
3. Patients receiving therapeutic doses of warfarin or heparin
4. Severe end organ disease
5. Patients who otherwise would not be candidates for radical prostatectomy because of health or tumour factors
6. Patients will be excluded if they had any prior malignancy unless the prior malignancy was diagnosed and definitively treated at least five years previously and there has never been any evidence of recurrence.
7. Other serious illness, psychiatric, or medical condition that would not permit the patient to be managed according to the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2008-05-13 (Actual); Study Completion 2008-05-13 (Actual)

PRIMARY OUTCOMES:
To assess the effects of combined neoadjuvant hormone therapy (NHT) and OGX-011 prior to radical prostatectomy on pathologic complete response rates in men with high risk localized prostate cancer | See Detailed Description, Treatment Plan

SECONDARY OUTCOMES:
To quantify changes in clusterin expression in residual prostate cancer after treatment with NHT and OGX-011 | See Detailed Description, Treatment Plan
To measure levels of full length OGX-011 in prostate tissues after 3 months of NHT | See Detailed Description, Treatment Plan
To assess the safety and tolerability toxicity of 3 months of OGX-011 and NHT prior to radical prostatectomy | See Detailed Description, Treatment Plan
To measure evidence of OGX-011's effect on clusterin expression in patient peripheral blood mononuclear cells (PBMNC) | See Detailed Description, Treatment Plan
To measure evidence of OGX-011's effect on patient clusterin serum levels | See Detailed Description, Treatment Plan
To assess the effects of combined NHT and OGX-011 on time to prostate specific antigen (PSA) nadir | See Detailed Description, Treatment Plan
To determine PSA recurrence rates after combined NHT and OGX-011 | See Detailed Description, Treatment Plan

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kim Chi, Principal Investigator — University of British Columbia
Locations (1):
- BC Cancer Agency and Vancouver General Hospital, Vancouver, British Columbia, Canada